CLINICAL TRIAL: NCT05605184
Title: Eine Anonyme Umfrage Bei Brustkrebspatient*innen Zum Thema Nutzerverhalten Von Gesundheits-Apps
Brief Title: Anonymous Survey of Breast Cancer Patients Concerning Their Use of Medical Apps
Acronym: Survey_App
Status: Active, not recruiting | Type: Observational
Sponsor: Technical University of Munich (Other)
Responsible Party: Principal Investigator, Heike Jansen, Principal Investigator, Technical University of Munich
Other Study IDs: Survey_App
Record Dates: First submitted 2022-08-12; First posted 2022-11-04 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Health Care Survey
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Survey: Breast cancer patients complete questionnaire concerning their use of medical apps.
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — Survey

SUMMARY:
Breast cancer patients complete questionnaires concerning their use of medical apps.

DETAILED DESCRIPTION:
Breast cancer patients of the department of gynecology at Technical University of Munich and Berlin Charité complete quesionnaires during routine appointments. Intention of the survey is to evaluate the importance of medical apps and the special needs of breast cancer patients. Moreover approaches to improve health care of breast cancer patients are expected to be developed.

ELIGIBILITY:
Inclusion Criteria:

* breast cancer patients
* patients who are legally competent and able to understand and follow instructions of the study staff

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Breast cancer patients at TUM Department of Gynecology and Obstetrics
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
The attitudes of breast cancer patients regarding the use of medical apps: a survey-based study | 6 Months
  Evaluation of relative frequency of answers in the questionnaire regarding patient's approach to app-utility

CONTACTS AND LOCATIONS:
Overall Officials: Heike Jansen, Dr. med., Principal Investigator — Technical University of Munich
Locations (1):
- Klinikum rechts der Isar, Frauenklinik, Technische Universität München, Munich, Germany, Germany

IPD SHARING:
Plan to Share IPD: No